CLINICAL TRIAL: NCT00480844
Title: Comparison of Cognitive Functions of Schizophrenic Patients Treated With Sertindole Versus Risperidone
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Prof. Mark Weiser, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-07-4639-JL-CTIL
Record Dates: First submitted 2007-05-30; First posted 2007-05-31 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Schizophrenia
Keywords: schizophrenia; Sertindole; Risperidone; cognitive impairment
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction | interventions — sertindole; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sertindole (Experimental)
  Interventions: Drug: Sertindole
- Risperidone (Active Comparator)
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Sertindole — Oral (tablets), 16-24 mg QD (once a day) for 12 weeks.
  Other Names: Serdolect
  Arms: Sertindole
Drug: Risperidone — Oral (tablets), 4-8 mg QD (once a day) for 12 weeks.
  Other Names: Rispond; Risperdal; Risperidex
  Arms: Risperidone

SUMMARY:
In this study we intend to compare the effect of Sertindole to that of Risperidone on cognitive impairment in schizophrenia.

Hypothesis: Sertindole will be as effective as Risperidone for treating cognitive impairment in schizophrenia and with fewer side effects.

DETAILED DESCRIPTION:
Introduction:

In this proposal we intend to compare the effect of Sertindole to that of Risperidone on cognitive impairment in schizophrenia.

Hypothesis:

Sertindole will be as effective as Risperidone for treating cognitive impairment in schizophrenia and with fewer side effects.

Study Drugs:

Risperidone is an "atypical" antipsychotic drug, being used widely all over the world. In Israel, Risperidone has been the first line drug for schizophrenia at the past decade. This drug was shown to be efficacious with bearable side effects. The side effects include: tiredness, dizziness, muscle dystonia, increased appetite and weight, dry mouth, constipation, tremor, orthostatic hypotension.

Sertindole is another "atypical" antipsychotic drug. The drug has been approved by the Israeli Ministry of Health. Sertindole was initially marketed in Britain on 1996. It was taken off the market, following several reports of cardiovascular deaths suspected to be caused by the drug (i.e. prolongation of the QT-interval in the ECG, suspected to cause ventricular arrhythmias). After renewing research, investigating more then 10000 patients for several years, the drug was found to be as safe as other antipsychotics. On 2002, the European union decided to put the Sertindole to the market.

Common Sertindole side effects are: dizziness, parasthesias, edema, orthostatic hypotension, nasal congestion, dyspnea, dry mouth, decreased semen volume, increased weight, prolongation of QT-interval in ECG.

Subjects and methods:

Overview: We propose to perform a multi-center, randomized, parallel-group, open-label study administering Sertindole or Risperidone to patients with schizophrenia, N=60. The primary outcome measure will be cognitive functioning. Secondary outcome measures will be discontinuation due to all causes, symptomatology and adverse events.

Procedure and Instruments:

Subjects:

Sixty male and female subjects will be recruited from patients treated in the inpatient and outpatient units in the Department of Psychiatry of the Sheba Medical Center, the Beer-Yaakov Mental Health Center and the Kfar Shaul Mental Health Center. Before inclusion into the study, patients will receive a careful medical workup, including complete medical history, physical examination; routine blood chemistry and blood count, EKG and urinalysis.

Inclusion and exclusion criteria will be based on the SmPCs of both compounds.

Medication:

The doses of study medication used will be based on the doses currently recommended by the manufacturers: Sertindole: 16-20 mg/day (in exceptional cases subjects will receive 24 mg/day, based on the clinical reasoning) or Risperidone 4-8 mg/day.

Duration:

Duration of randomized, open-label treatment will be 12 weeks. Following this phase, an additional 12 week phase with Sertindole will be offered to subjects who were previously randomized to the Risperidone arm.. As per IRB requirements, patients responding to Sertindole will be eligible to receive Sertindole as compassionate care(in accordance wit MOH requirements for compassionate care)

Assessment instruments:

* the following assessment scales will be administered before randomization, after 12 weeks of randomized treatment, and , if applicable, following 12 weeks of with Sertindole Positive symptoms will be assessed by PANSS (Positive and Negative Syndrome Scale)
* Negative symptoms will be assessed by SANS (Scale of the Assessment of Negative Symptoms)
* Cognitive functioning will be assessed using MATRICS (Measurement And Treatment Research to Improve Cognition in Schizophrenia).
* Movement disorders will be assessed by the Simpson Angus Scale and AIMS (Abnormal Involuntary Movement Scale) scales
* Blood levels of glucose, triglycerides and cholesterol
* Weight, height, and vital signs will be measured and recorded
* ECG

Tests which are language-sensitive have been standardized and will be in assessed in Hebrew. Assessment will be made by a rater who is blinded to the treatment.

Concomitant Medications:

Patients receiving mood-stabilizers, anti-depressants, sedatives and hypnotics will be allowed to participate in the study only if they are on a stable dose of these medications for 2 weeks before entering the trial. After randomization, changes in the doses of concomitant medications will be recorded and analyzed at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from Schizophrenia (DSM IV).
* Failure of at least one previous antipsychotic for intolerance.
* Psychotic symptoms that are not secondary to a general medical condition or substance abuse.
* Ages between 18-65 years old.
* Patients receiving other psychotropic medications (anti-depressants, mood stabilizers, sedatives, hypnotics) must be on a stable dose for at least 2 weeks before entering the trial.
* Able to understand and sign an informed consent form.

Exclusion Criteria:

* Patients suffering from psychotic disorders caused by a general medical condition.
* Patients having high suicidal risk, as measured by score of 2 or more in CDSS - Calgary Depression Scale for Schizophrenia.
* Patients suffering from an unstable clinically significant medical condition (endocrine, nutritional, hepatic, urinary).
* Significant cardiovascular illness, and/or QT prolongation at screening (more then 450 msec for male or 470 msec for female).
* Patients suffering from a malignancy or neuro-degenerative illness (e.g. Parkinsons' Disease)
* Patients suffering from organic brain disorders, including epilepsy and mental retardation.
* Patients suffering from a clinically significant mood disorder.
* Pregnancy.
* History of drug or alcohol dependence within the last year.
* Previous documented non-response to Risperidone.
* Patients using medicinal products that are contraindicated with sertindole and/or Risperidone.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-10; Primary Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
cognitive functioning | 24 weeks

SECONDARY OUTCOMES:
Discontinuation due to all causes, symptomatology and adverse events. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark Weiser, Dr, Principal Investigator — Shaba Medical Center, Tel-Aviv University Sackler School of Medicine
Locations (3):
- Israel (3):
  - Department of Psychiatry of the Sheba Medical Center, Ramat Gan, Tel Hashomer
  - Beer-Yaakov Mental Health Center, Beer-Yaakov
  - Kfar Shaul Mental Health Center, Jerusalem